CLINICAL TRIAL: NCT01683422
Title: A Phase II Trial of Gemcitabine and Erlotinib (GE) Plus Proton-chemotherapy (PCT) and Capox for Locally Advanced Pancreatic Cancer (LAPC)
Brief Title: Chemotherapy Plus Proton-chemotherapy for Locally Advanced Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Updated chemotherapy regimens currently evaluated in clinical trials due to lack of progress in treating this condition; analysis continues in the realm of patterns of failure and increasing quality of life
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gary Yang, MD, MD, Principal Investigator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5110324
Record Dates: First submitted 2012-02-17; First posted 2012-09-11 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Protons; Gemcitabine; Erlotinib Hydrochloride; Capecitabine; Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Proton Radiation (Experimental): Pre-Proton-chemotherapy (PCT) Patients will receive a combination of the agents (Gemcitabine plus Erlotinib) for 8 weeks prior to PCT Gemcitabine 1000 mg/m2 IV, days 1, 8, 15, 29, 36 and 43 Erlotinib 100 mg po qd days 1-43
  PCT to be started in 4 to 8 weeks after completion of Pre-PCT Proton therapy: 50.4 Gy/28 fractions (1.8 Gy per fraction) once a day for 5 ½ weeks.
  Chemotherapy: Capecitabine 825mg/m2 po bid M-F, starting on day 1 of proton therapy until proton therapy completed
  Post-PCT to be started in 4 to 6 weeks after completion of PCT Oxaliplatin 130 mg/m2, day 1 Capecitabine 1000 mg/m2 po bid on days 2 to 15 for 14 days The CapOx regimen (Capecitabine plus Oxaliplatin) is repeated every 3 weeks for 4 cycles
  Interventions: Radiation: Proton, Gemcitabine, Erlotinib, Capecitabine; Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Proton, Gemcitabine, Erlotinib, Capecitabine — Gemcitabine 1000 mg/m2 iv, days 1, 8, 15, 29, 36 and 43 Erlotinib 100 mg po qd days 1-43 Capecitabine 825mg/m2 po bid M-F, starting on day 1 of proton therapy until proton therapy completed.
  Post-proton chemotherapy: To be started in 4 to 6 weeks after completion of proton chemotherapy. Oxaliplatin 130 mg/m2 po bid on days 2 to 15 for 14 days. The CapOx regimen (Capcitabine plus Oxaliplatin) is repeated every 3 weeks for 4 cycles.
Radiation: Proton Radiation

SUMMARY:
The current trial will provide important data on the recurrence rates and patterns of failure using state of the art target agent, chemotherapy and proton beam technology for patients with Locally Advanced Pancreatic Cancer (LAPC). A median survival of 10 months or greater would be considered evidence of a regimen potentially worthy of further study as a new treatment paradigm in one arm in a future phase III trial.

DETAILED DESCRIPTION:
The current trend toward using the biology of the disease as it becomes evident over a period of chemotherapy to better select patients who will benefit from chemoradiotherapy (CRT) seems to be the most pragmatic way to proceed, until we have a better means of predicting tumor behavior and more active systemic agents. This has led to increased interest in treatment regimens incorporating induction chemotherapy with target agent followed by CRT and additional chemotherapy for diseases that carry a high risk for systemic relapse.

The PA.3 trial was the first phase III trial in advanced pancreatic cancer to show a survival advantage with the addition of a second drug, in this case the oral Epidermal growth factor receptor (EGFR) inhibitor Erlotinib to gemcitabine. The approval provides an important proof of concept regarding the use of newer "targeted" therapies in pancreatic cancer 7. Proton beam therapy may result in lower toxicity, enhanced efficacy and could contribute to improved local control of patients with LAPC. The capecitabine and oxaliplatin ((CapOx)) regimen utilized in this trial has been proven to be active in gemcitabine-pretreated patients with advanced pancreatic cancer.

The current trial will provide important data on the recurrence rates and patterns of failure using state of the art target agent, chemotherapy and proton beam technology for patients with LPAC. A median survival of 10 months or greater would be considered evidence of a regimen potentially worthy of further study as a new treatment paradigm in one arm in a future phase III trial.

Patients with unresectable or borderline resectable non-metastatic adenocarcinoma of the pancreas, as defined by 2012 National Comprehensive Cancer Network (NCCN) guidelines, were included. Patients received neoadjuvant gemcitabine 1000 mg/m2 IV on days 1, 8, 15, 22, 29, 36, and 43 and erlotinib 100 mg by mouth every day for 1-43 days (GE). If there was no evidence of metastatic disease after GE, then patients preceded with proton therapy to 50.4 Gy in 28 fractions with concurrent capecitabine 825 mg/m2 twice per day (PCT). This was followed with maintenance oxaliplatin 130 mg/m2 on day 1 and capecitabine 1000 mg/m2 twice per day on days 2 to 15 (CapOx) for 4 cycles. The primary study objective was 1-year overall survival (OS). The benchmark was 43% 1-year survival as demonstrated in Radiation Therapy Oncology Group (RTOG/NRG) 98- 12. The Kaplan-Meier method was used to estimate the one-year OS and the median OS and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable non-metastatic adenocarcinoma of the pancreas
* The American Joint Committee on Cancer (AJCC) stage I-III with unresectable or borderline unresectable disease as defined by NCCN guidelines
* Radiological resectability is defined by the following criteria on abdominal imaging:

  1. No evidence of tumor extension to the celiac axis, hepatic artery or superior mesenteric artery.
  2. No evidence of tumor encasement or occlusion of the superior mesenteric vein (SMV) or the SMV/portal vein confluence
  3. No evidence of visceral or peritoneal metastases
* Borderline and Unresectable cases would be defined as those that do not meet the criteria in section and also show no evidence of distant metastatic or intraperitoneal disease.
* Eastern Cooperative Oncology Group performance status of ≤ 2
* Age > 18 years
* Adequate hematologic reserve, hepatic reserve and renal function
* White Blood Cell (WBC) > 2,000 cells/mm3
* Absolute Neutrophil Count (ANC) > 1,500 cells/mm3
* Platelets > 100,000 cells/mm3
* Serum bilirubin ≤ 2.5 mg/dL
* Serum creatinine ≤ 2 x upper limit of normal (ULN), or creatinine clearance (Ccr) ≥ 30ml/min
* Alanine aminotransferase (ALT) < 3 times ULN
* Aspartate transaminase (AST) < 3 times ULN
* Albumin > 3.2 g/dl
* Patient must sign study-specific informed consent

Exclusion Criteria:

* AJCC stage IV with metastatic disease
* Eastern Cooperative Oncology Group performance status of > 2
* Age < 18 years
* WBC < 2,000 cells/mm3
* ANC < 1,500 cells/mm3
* Platelets > 100,000 cells/mm3
* Serum bilirubin > 2.5 mg/dL
* Serum creatinine > 2 x upper limit of normal (ULN), or creatinine clearance (Ccr) ≥ 30ml/min
* ALT > 3 times ULN
* AST > 3 times ULN
* Albumin < 3.2 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Yang, MD, Principal Investigator — gyang@llu.edu
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanghvi SM, Coffman AR, Hsueh CT, Kang J, Park A, Solomon NL, Garberoglio CA, Reeves ME, Slater JD, Yang GY. A phase II trial of gemcitabine and erlotinib followed by ChemoProton therapy plus capecitabine and oxaliplatin for locally advanced pancreatic cancer. J Gastrointest Oncol. 2022 Aug;13(4):1989-1996. doi: 10.21037/jgo-22-327. PMID 36092320

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton Radiation: Proton, Gemcitabine, Erlotinib, Capecitabine: Gemcitabine 1000 mg/m2 iv, days 1, 8, 15, 29, 36 and 43 Erlotinib 100 mg po qd days 1-43 Capecitabine 825mg/m2 po bid M-F, starting on day 1 of proton therapy until proton therapy completed.
  Post-proton chemotherapy: To be started in 4 to 6 weeks after completion of proton chemotherapy. Oxaliplatin 130 mg/m2 po bid on days 2 to 15 for 14 days. The CapOx regimen (Capcitabine plus Oxaliplatin) is repeated every 3 weeks for 4 cycles.
  Proton Radiation
Period: Overall Study
Arm/Group | Proton Radiation
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Proton Radiation: Radiation: Proton, Gemcitabine, Erlotinib, Capecitabine Gemcitabine 1000 mg/m2 iv, days 1, 8, 15, 29, 36 and 43 Erlotinib 100 mg po qd days 1-43 Capecitabine 825mg/m2 po bid M-F, starting on day 1 of proton therapy until proton therapy completed.
  Post-proton chemotherapy: To be started in 4 to 6 weeks after completion of proton chemotherapy. Oxaliplatin 130 mg/m2 po bid on days 2 to 15 for 14 days. The CapOx regimen (Capcitabine plus Oxaliplatin) is repeated every 3 weeks for 4 cycles.
  Radiation: Proton Radiation
Arm/Group | Proton Radiation
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 59.6 [47 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 2
  Unknown or Not Reported | 1
Proton Radiation [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: One-year Survival Rate
Description: Subjects will be followed after treatment completed to determine length of survival rate. The primary study objective was 1-year overall survival (OS, failure: death due to any cause). The Kaplan-Meier method was used to estimate the one-year OS. Secondary Objectives were the frequency of serious adverse events, disease control rate and progression-free survival.
Time Frame: One year after treatment completed.
Population: The study enrolled 9 patients between January 2013 and March 2016, when the trial was closed due to poor accrual.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 9
percentage of participants | 55.6 [31 to 99]
Statistical Analysis 1: Comparison: Proton Radiation; In the RTOG 9812 (NCT00003591) for unresectable pancreatic cancer, a one-year survival rate of 43% was observed. There were 109 analyzable patients on NCT00003591 with 61 still at risk for death at one year. Using the method of Dixon and Simon, a sample size of 39 analyzable patients followed over 12 months will ensure at least 90% probability of detecting a minimum of 17% improvement in the one-year survival rate compared to NCT00003591 at the 0.10 significance level (with a one-sided test); Test type: Superiority — The reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; p = 0.1, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 years
Description: Patients with locally advanced pancreatic cancer--9 patients died due to recurrence of disease. Entered as serious Adverse Event (AE)
Groups:
- Proton Radiation: Gemcitabine 1000 mg/m2 iv, days 1, 8, 15, 29, 36 and 43 Erlotinib 100 mg po qd days 1-43 Capecitabine 825mg/m2 po bid M-F, starting on day 1 of proton therapy until proton therapy completed.
  Post-proton chemotherapy: To be started in 4 to 6 weeks after completion of proton chemotherapy. Oxaliplatin 130 mg/m2 po bid on days 2 to 15 for 14 days. The CapOx regimen (Capcitabine plus Oxaliplatin) is repeated every 3 weeks for 4 cycles.
Arm/Group | Proton Radiation
All-Cause Mortality (participants affected / at risk) | 9/9
Serious Adverse Events (participants affected / at risk) | 9/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation (N=9)
serious (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) — metastatic disease

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-09-27): https://cdn.clinicaltrials.gov/large-docs/22/NCT01683422/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT01683422/ICF_001.pdf